CLINICAL TRIAL: NCT00520260
Title: Bromfenac 0.09% vs. Ketorolac 0.4% During the Induction Phase of Treatment With Topical Cyclosporine for Chronic Dry Eye Patients
Brief Title: Bromfenac 0.09% vs Ketorolac 0.4% for Cyclosporine Induction Phase
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Florida Eye Microsurgical Institute (Other)
Collaborators: Bausch & Lomb Incorporated (Industry)
Responsible Party: Barry Schechter, MD, Florida Eye Microsurgical Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Sch012007
Record Dates: First submitted 2007-08-21; First posted 2007-08-23 (Estimated); Last update posted 2009-02-19 (Estimated); Status verified 2009-02

CONDITIONS: Dry Eye Disease; Ocular Comfort
MeSH Terms: conditions — Dry Eye Syndromes | interventions — bromfenac; Ketorolac

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Active treatment arm bromfenac 0.09% BID for 6 weeks
  Interventions: Drug: bromfenac
- 2 (Active Comparator): ketorolac 0.4% BID for 6 weeks
  Interventions: Drug: ketorolac

INTERVENTIONS:
Drug: bromfenac — 0.09%, BID, 6 weeks
  Arms: 1
Drug: ketorolac — 0.4%, BID, 6 weeks
  Arms: 2

SUMMARY:
To compare bromfenac 0.09% and ketorolac 0.4% when used concomitantly with cyclosporine ophthalmic emulsion 0.05% in improving patient comfort during the induction phase of treatment for chronic dry eye disease

ELIGIBILITY:
Inclusion Criteria:

* Must be in general good health
* Diagnosis of moderate to severe dry eye syndrome

Exclusion Criteria:

* Patients who are unlikely to respond to cyclosporine ophthalmic emulsion therapy
* Patients who are pregnant or nursing females
* Unwilling to discontinue use of contact lenses during the run-in and duration of the study
* Presence or history of any systemic or ocular disorder or condition that could possibly interfere with the interpretation of the study results in the study eye
* Previous treatment failure on CSA 0.05% (Restasis)
* Known hypersensitivity to any component of the study or procedural medications
* Participation in any other clinical trial within 30 days prior to screening
* Known contraindication to any study medication or any of their components.
* Should not be taking any oral anti-histamines, beta blockers or diuretics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2007-08; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Ocular comfort | six weeks

CONTACTS AND LOCATIONS:
Overall Officials: Barry Schechter, MD, Principal Investigator — Florida Eye Microsurgical Institute
Locations (1):
- Florida Eye Microsurgical Institute, Boynton Beach, Florida, United States